CLINICAL TRIAL: NCT06574061
Title: Evaluation in Routine Practice of the Benefits of Sublingual Allergen Immunotherapy in Allergic Patients According to Different Modalities of Use
Brief Title: Evaluation of the Benefits of Sublingual AIT (PRACTIS)
Acronym: PRACTIS
Status: Completed | Type: Observational
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Other Study IDs: OTH-PES-08-FR
Record Dates: First submitted 2024-08-01; First posted 2024-08-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Allergic Rhinitis
Keywords: SLIT treatment, patient adherence/satisfaction, PBI
MeSH Terms: conditions — Rhinitis, Allergic; Patient Compliance; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study was to evaluate in routine practice the benefits of sublingual allergen immunotherapy (SLIT) for allergic patients with allergic rhinitis (AR), with or without asthma, according to various methods of use (treatment regimen: formulation type, dose, duration, initiation) and type of allergen (grass pollen, tree pollen, herbaceous pollen, house dust mites, animal dander, moulds and poly-reactive types).

DETAILED DESCRIPTION:
The treatment considered was any SLIT (tablet or liquid forms) accepted by the patient and the parent(s) in the case of minor patients. The treatment was taken as prescribed by the observing physician.

The expected benefits for patients after approximately 6 and 12 months after initiation of SLIT included:

* Decreased intensity of symptoms
* Decreased discomfort
* Decreased consumption of symptomatic treatments or associated treatments (especially in asthmatic patients)
* Improved quality of life
* Reduced absenteeism from school or work
* Beneficial impact on leisure activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 years or older
* Patients with a respiratory allergy with significant clinical symptoms and whose diagnosis was confirmed by a positive skin prick-test and/or the presence of specific IgE antibodies to one or more allergens implicated in the symptoms
* Patients eligible for AIT (patients who had been treated with AIT in the 3 years prior to the inclusion visit could be included if starting a new form and/or type of AIT)
* Patients previously treated with a pharmacological AR treatment in the month before the inclusion visit or during the previous pollen season, and requiring the initiation of AIT
* Patients (and/or their parents or legal representatives as appropriate) agreeing to take part in the study after having been informed orally and in writing by the observing physician.

Exclusion Criteria:

* Patient with a hypersensitivity (allergy) to any of the excipients in the selected AIT
* Patients taking beta-blockers (including local treatments, e.g. eye drops)
* If asthmatic patient:
* Patients with uncontrolled (unstable) or severe asthma (in adults this was defined as daily symptoms and FEV1 <70% of the theoretical value after appropriate drug treatment, and in children and adolescents by FEV1 <80% of the theoretical value after appropriate drug treatment)
* Patients who have had a severe asthma exacerbation in the last three months
* Asthmatic patient with unresolved acute infection of the airways.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population included adult patients, adolescents and children (aged ≥5 years) with an allergy to one or more allergens confirmed by a positive skin prick-test and/or the presence of specific IgE antibodies, and eligible for AIT.
Sampling Method: Probability Sample
Enrollment: 1635 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
PBQ (Patient Benefit Questionnaire) | V1 / V2 (6, 9 or 12 months after treatment initiation)
  The Patient Benefit Questionnaire (PBQ) was used as the primary endpoint to evaluate the benefits perceived by patients.

SECONDARY OUTCOMES:
PNQ (Patient Need Questionnaire) | V1 (at study inclusion)
  The Patient Need Questionnaire (PNQ) was used to evaluate the expectations of patients regarding the prescription or new treatment(s) prescribed by the observing physicians.
PBI Patient Benefit Index | Patient self-questionnaires returned at V1 (at study inclusion) and V2 (6, 9 or 12 months after treatment initiation)
  The overall PBI score was calculated using the PNQ questionnaire at V1 (treatment expectations) and the PBQ questionnaire at V2 (treatment benefits).
  PBI is an index of the benefits perceived by patients with the AIT received. It considers patient expectations prior to AIT treatment and the perceived benefits after treatment.
  A PBI ≥1 is considered as indicating a relevant benefit of the AIT treatment for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, Professor, Principal Investigator — CHU & IDESP, Montpellier, France
Locations (1):
- Stallergenes Greer, Antony, France

IPD SHARING:
Plan to Share IPD: No